CLINICAL TRIAL: NCT03543254
Title: "Follow the Sutures". An Open Multicenter, Multinational Pilot Study to Explore Tolerability, Safety and Effect of a New Procedure for Injecting Botulinum Toxin in the Head Against Chronic Migraine
Brief Title: "Follow the Sutures". A New Procedure for Injection of Botulinum Toxin for Chronic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1490; 2017-002516-13 (EudraCT Number)
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Migraine Disorders; Chronic Disease
Keywords: Botulinum Toxins, Type A; Injections; Cranial Sutures; Head
MeSH Terms: conditions — Migraine Disorders; Chronic Disease | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BoNT-A injected (Experimental): BoNT-A (Botulinum toxin A) injected in the head on specific sites and in half the usual concentration
  Interventions: Drug: BoNT-A

INTERVENTIONS:
Drug: BoNT-A — 90U BoNT-A, given in one treatment as 18 injections of 5u (0.2 ml) each, on specific preselected sites along the sutures of the skull.
  First 100 U of Botox® is solved in 4 ml (cc) of isotone saline water (9 mg/ml), distributed in 4 syringes. This is half the usual concentration, allowing for better diffusion in order to reach the target structures.
  Other Names: Botox; Botulinum Toxin Type A

SUMMARY:
There is no doubt that chronic migraine is a large public health problem, which is both disabling and costly. Many patients and headache doctors see Botulinum toxin (Botox) treatment as a big stride forward, but it is a problem that the effect has been shown in only one study, with a low therapeutic gain. For this reason, before this costly treatment is expanded to potentially several thousand patients in Norway, it would be highly desirable that 1) there is additional good scientific evidence for use of Botox , 2) a more effective treatment procedure is developed, 3) the potential for unblinding is reduced, and 4) the dose, number of injection sites and cost can be halved, and 5) the adverse effects are minimized. These may be the results of this pilot project where injections are given along the sutures, which can open up for a later randomized, blinded and controlled study.

DETAILED DESCRIPTION:
The study is an an open-label, non-con trolled, single-arm and single-center phase II study, at the outpatient clinic of the Department of Neurology and Clinical neurophysiology at St. Olavs Hospital, Trondheim, Norway. The study was originally also planned at the Mayo Clinic, Scottsdale, AZ, USA, but because the study there had not been started before the COVID-19 pandemic, the study was performed only in Trondheim. Potential study participants should be identified among the regular outpatients at the Department of Neurology at St. Olavs hospital. Potential participants should recceive an email with the informed consent form, which should be signed at the screening visit where a detailed medical history and medical examination should be per formed. Patients should complete a paper head ache diary, recording pain intensity and duration, concomitant migraine symptoms (nausea, vomiting, phono- and photophobia), acute medication (type, number of doses) and work absence (yes/no/not relevant). Also, they should record any adverse events. After 7-14 days, they should receive a telephone call from a nurse asking about adverse events and concom itant medication and reminding them to maintain the daily diary. After a baseline period of at least 28 days, diaries should be reviewed at a treatment visit, and each participant should receive injections according to the described procedure. Women of child bearing potential should have a negative pregnancy test before the injections. The duration of the injection procedure should be measure with a stopwatch and immediately after the injections, the patient should be asked to record on a VAS scale (0-10) the level of pain of the procedure and the investigator recorded the degree of bleeding (no, mild, moderate, marked) and any other injection-related adverse events (AEs). Patients should then be asked were asked to keep a headache diary for another 12 weeks or more, before the end of the study visit. During this period, they should receive a call from the study nurse at weeks 2 and 9, reminding to keep the headache diary, and asking about AEs and concomitant medication. They should be also asked whether they had noticed any change in their ability to make forehead wrinkles (no, little, moderate, marked, full paralysis)

ELIGIBILITY:
Inclusion Criteria:

* Chronic migraine, as defined in the ICHD-3 beta version
* Chronic migraine should have been present for at least ½ year prior to evaluation for study inclusion
* For women of child-bearing potential there must be no pregnancy or planned pregnancy during the study period, and use of highly effective contraception
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations

Exclusion Criteria:

* Diseases that are contraindications for use of Botulinum toxin A (Myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, other diseases interfering with neuromuscular function)
* Allergy to Botulinum toxin A
* Other primary or secondary headache disorder, including medication overuse headache (MOH). This means that at least one attempt to withdraw acute medication should have been performed earlier, but without success
* Severe depression or other psychiatric disorder that may interfere with the treatment
* Abuse of alcohol or illicit drugs
* Use of more than one headache prophylactic medication, or change in type and dose of prophylactic medication < 28 days before start of baseline period
* Previous exposure at any time to any botulinum toxin serotype
* Infection at one or more injection site(s)
* Having received extracranial nerve block, cervical facet injection, or other interventional procedure for headache within the prior 3 months
* Use of opioids or barbiturate containing medication(s) > 10 days per month within the preceding 3 months
* Participating in another trial that might affect the current study
* Should not participate in the opinion of the investigator (e.g. not able to comply with study procedures).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geir Bråthen, md, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No
No plans

REFERENCES:
- [Derived] Stovner LJ, Hagen K, Tronvik E, Bruvik Gravdahl G, Burstein R, Dodick DW. FollowTheSutures: Piloting a new way to administer onabotulinumtoxinA for chronic migraine. Cephalalgia. 2022 Jun;42(7):590-597. doi: 10.1177/03331024211067775. Epub 2022 Feb 15. PMID 35166150
- See also: Published paper in Cehalalgia — https://pubmed.ncbi.nlm.nih.gov/35166150/

RESULTS

PARTICIPANT FLOW:
Groups:
- BoNT-A Injected: BoNT-A (Botulinum toxin A) injected in the head on specific sites and in half the usual concentration
  BoNT-A: 90U BoNT-A, given in one treatment as 18 injections of 5u (0.2 ml) each, on specific preselected sites along the sutures of the skull.
  First 100 U of Botox® is solved in 4 ml (cc) of isotone saline water (9 mg/ml), distributed in 4 syringes. This is half the usual concentration, allowing for better diffusion in order to reach the target structures.
Period: Overall Study
Arm/Group | BoNT-A Injected
Started | 20
Completed | 19 (The last patient being lost to follow up after the baseline period)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: 20 patients with chronic migraine
Arm/Group | BoNT-A Injected
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: adverse events (other than clearly related to migraine) will be recorded in the diary by the patients and reviewed during the scheduled visits
Time Frame: 12 weeks
Population: All included got injection of botulinum toxin. One out of 19 (5.3%) had reduced power of chewing
Measure: Count of Participants; unit: Participants
Arm/Group | BoNT-A Injected
Number analyzed (Participants) | 19
Participants | 1

2. Secondary Outcome: Injection Time
Description: Time used for injection of Medicine measured by stopwatch
Time Frame: Week 1
Population: Time used for injection of Medicine measured by stopwatch (not measured in 3 patients)
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- BoNT-A Injection: 19 patents received botulinum-toxin, and time used to injection measured by stopwatch in 16 patients
Arm/Group | BoNT-A Injection
Number analyzed (Participants) | 16
Minutes | 5.47 (1.02)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events (serious and not serious)
Arm/Group | BoNT-A Injected
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BoNT-A Injected (N=19)
Power of chewing (Musculoskeletal and connective tissue disorders) | 1 (1) — Reduced power of chewing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT03543254/Prot_002.pdf
  • Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT03543254/SAP_003.pdf
  • Informed Consent Form (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT03543254/ICF_004.pdf